CLINICAL TRIAL: NCT07148063
Title: Association of Preoperative Inflammatory Biomarkers With Postoperative Nausea and Vomiting in Children Undergoing Orchiopexy
Brief Title: Inflammatory Biomarkers as Predictors of PONV Following Pediatric Orchiopexy
Status: Recruiting | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Sule Ozdemir, Principal İnvestigator, Ankara Etlik City Hospital
Other Study IDs: AEŞH-EK-2025-205
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Anesthesia; Postoperative Nausea and Vomiting (PONV); Inflammatory Biomarkers
Keywords: Pediatric anesthesia; Orchiopexy; Postoperative Nausea and Vomiting (PONV); Inflammatory biomarkers
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measurement of Preoperative Inflammatory Biomarkers — Blood samples will be collected preoperatively to measure inflammatory biomarkers, including neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), systemic immune-inflammation index, monocyte-to-lymphocyte ratio (MLR), and systemic inflammation response index. These values will be analysed in relation to the incidence of postoperative nausea and vomiting within the first 6 hours after pediatric orchiopexy. No experimental drug or device will be administered as part of the study; all procedures will be conducted within the scope of standard perioperative care.

SUMMARY:
Orchiopexy is a common surgical procedure for the treatment of cryptorchidism in the pediatric population, with a high incidence of postoperative nausea and vomiting (PONV).

Recent evidence suggests that systemic inflammation may contribute to PONV pathogenesis, and preoperative inflammatory biomarkers such as NLR, PLR, SII, MLR, and SIRI could serve as predictive indicators.

This prospective observational study aims to evaluate the relationship between these biomarkers and PONV incidence in children undergoing orchiopexy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 1 and 8 years
* Patients with ASA physical status I-II
* Patients scheduled for elective orchiopexy
* Obtained written informed consent from parents/guardians

Exclusion Criteria:

* Patients younger than 1 year or older than 8 years
* Patients with ASA physical status III or higher
* Presence of acute infection signs
* History of previous nausea or vomiting

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1-8 years with ASA physical status I-II who are scheduled to undergo elective orchiopexy under general anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-03-13 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Nausea and Vomiting (PONV) | Within 6 hours postoperatively
  PONV will be assessed using a standardized nausea-vomiting scoring system by an anesthesiologist blinded to biomarker results.

SECONDARY OUTCOMES:
Need for Antiemetic Treatment | Within 6 hours postoperatively
  The number of patients who receive at least one dose of rescue antiemetic medication will be recorded within the first 6 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Altındağ, Ankara, Turkey (Türkiye)